CLINICAL TRIAL: NCT01707316
Title: A Double-Blind, Randomized, Placebo-Controlled, 3-Way Cross-Over Study to Evaluate the Single-Dose Pharmacokinetics and Pharmacodynamics of JNJ-28431754 (Canagliflozin) in Healthy Chinese Subjects
Brief Title: A Study to Assess the Pharmacokinetics and Pharmacodynamics of Canagliflozin in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR100923; 28431754DIA1026 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Healthy; JNJ-28431754; Canagliflozin; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1: Treatment A-B-C (Experimental): The study consists of 3 single-dose treatment periods. Each treatment period will be 5 days in duration. Successive treatment periods will be separated by a washout period (with no medication) of 10 days.
  Interventions: Drug: Treatment A: Canagliflozin 100 mg; Drug: Treatment B: Canagliflozin 300 mg; Other: Treatment C: Placebo
- Sequence 2: Treatment B-C-A (Experimental): The study consists of 3 single-dose treatment periods. Each treatment period will be 5 days in duration. Successive treatment periods will be separated by a washout period (with no medication) of 10 days.
  Interventions: Drug: Treatment A: Canagliflozin 100 mg; Drug: Treatment B: Canagliflozin 300 mg; Other: Treatment C: Placebo
- Sequence 3: Treatment C-A-B (Experimental): The study consists of 3 single-dose treatment periods. Each treatment period will be 5 days in duration. Successive treatment periods will be separated by a washout period (with no medication) of 10 days.
  Interventions: Drug: Treatment A: Canagliflozin 100 mg; Drug: Treatment B: Canagliflozin 300 mg; Other: Treatment C: Placebo

INTERVENTIONS:
Drug: Treatment A: Canagliflozin 100 mg — Volunteers will receive one 100 mg over-encapsulated tablet of canagliflozin as a single oral (by mouth) dose on Day 1.
  Other Names: JNJ-28431754
Drug: Treatment B: Canagliflozin 300 mg — Volunteers will receive one 300 mg over-encapsulated tablet of canagliflozin as a single oral dose on Day 1.
  Other Names: JNJ-28431754
Other: Treatment C: Placebo — Volunteers will receive one matching placebo (inactive medication) capsule as a single dose on Day 1.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (what the body does to the medication) and pharmacodynamics (the action of the medication on the body) of JNJ-28431754 (canagliflozin) and its main metabolites (break-down products) following 2 different doses of canagliflozin in healthy Chinese volunteers. Safety and tolerability of canagliflozin will also be assessed.

DETAILED DESCRIPTION:
This study will be a double-blind (neither the Investigator nor volunteer knows the assigned treatment), randomized (the treatment is assigned by chance), placebo-controlled (one of the study treatments is inactive), single-dose, 3-way cross over study (all volunteers will receive each of the 3 treatments but in a different order) in healthy Chinese volunteers. Volunteers will be assigned to 1 of 3 treatment sequence groups (ABC, BCA, or CAB). The treatment sequence will be decided by randomization. Treatment A will be a single oral (by mouth) dose of 100 mg of canagliflozin. Treatment B will be a single oral dose of 300 mg of canagliflozin. Treatment C will be a single oral dose of placebo (inactive medication). Each treatment will be given during a treatment period of 5 days duration; each treatment period will be separated by a washout period (a time period with no medication) of at least 10 days. Canagliflozin is currently being investigated for the treatment of type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must be non-smokers for at least 6 months before first study drug administration
* Volunteers must consume no more than 4 to 5 cups of coffee or tea or 8 cans of cola each day

Exclusion Criteria:

* History of or currently active illness considered to be clinically significant by the Investigator or any other illness that the Investigator considers should exclude the patient from the study or that could interfere with the interpretation of the study results
* Female volunteer is breast-feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin and its major metabolites following a single 100 mg and 300 mg dose | Up to Day 4
  Plasma concentrations of canagliflozin and its major metabolites will be used to determine pharmacokinetic parameters (measurements that explore what the body does to the drug) for canagliflozin and its major metabolites.
Urine concentrations of canagliflozin and its major metabolites following a single 100 mg and 300 mg dose | Up to Day 2
  Urine concentrations of canagliflozin and its major metabolites will be used to determine pharmacokinetic parameters for canagliflozin and its major metabolites.

SECONDARY OUTCOMES:
Renal threshold for glucose excretion following a single 100 mg dose of canagliflozin, 300 mg dose of canagliflozin, and placebo (inactive medication) | Up to Day 2
  Renal threshold is defined as the plasma glucose concentration above which glucose is excreted in the urine.
Urine glucose excretion (UGE) following a single 100 mg dose of canagliflozin, 300 mg dose of canagliflozin, and placebo (inactive medication) | Up to Day 2
  UGE is equal to the amount of glucose excreted into the urine over defined time intervals.
Mean plasma glucose concentration following a single 100 mg dose of canagliflozin, 300 mg dose of canagliflozin, and placebo (inactive medication) | Up to Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Beijing, China

REFERENCES:
- [Derived] Chen X, Hu P, Vaccaro N, Polidori D, Curtin CR, Stieltjes H, Sha S, Weiner S, Devineni D. Pharmacokinetics, Pharmacodynamics, and Safety of Single-Dose Canagliflozin in Healthy Chinese Subjects. Clin Ther. 2015 Jul 1;37(7):1483-1492.e1. doi: 10.1016/j.clinthera.2015.04.015. Epub 2015 Jun 3. PMID 26048186